CLINICAL TRIAL: NCT06271057
Title: Golcadomide (BMS-986369) Post-CAR T-cell in R/R Aggressive Large B-cell Lymphoma Patients With High Risk of Relapse
Brief Title: Golcadomide Post-CAR T-cell in R/R Aggressive Large B-cell Lymphoma Patients With High Risk of Relapse
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Lymphoma Study Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARMOD
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Diffuse Large B-cell Lymphoma Refractory; Refractory Primary Mediastinal Large B-Cell Lymphoma; Refractory Transformed B-cell Non-Hodgkin Lymphoma; Refractory High Grade B-Cell Lymphoma
Keywords: eligible for CAR T-cells therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- golcadomide post CAR T-cells (Experimental): 0.3 mg - Per Os - every week - 6 months
  Interventions: Drug: golcadomide

INTERVENTIONS:
Drug: golcadomide — golcadomide 0.3 mg weekly from D+5 post CAR T-cells administration until D+166
  Other Names: BMS-986369; CC-99282

SUMMARY:
This study is an open-label, multicenter, proof of concept, phase 2 trial. Patients will be recruited over 18 months. Safety analysis will be performed with a stop of the enrollment after 3 patients have either 1 complete treatment cycle or permanently discontinued treatment whichever occurs first.

Approximatively 65 patients with aggressive large B-cell lymphoma (LBCL) (including diffuse large B-cell lymphoma (DLBCL), Primary mediastinal B-cell lymphoma (PMBCL), any transformed follicular or marginal zone lymphoma, high-grade B-cell lymphoma (HGBL)) will be enrolled in the study.

The duration of treatment with golcadomide (CELMoD) is 24 weeks with 6 cycles of 28 days (4 weeks), starting at 5 days after CAR-T cells infusion.

The primary objective of the study is to estimate the efficacy of golcadomide administered post-anti-CD19 CAR T-cell infusion, Efficacy determination will be based upon the primary endpoint of complete metabolic response (CMR) rate at 3 months after infusion of anti-CD19 CAR T-cell assessed by study investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who understood and voluntarily signed and dated an informed consent prior to any study-specific assessments/procedures being conducted
2. Adults patients (≥ 18-year-old at the time of signing the informed consent form; no upper age limit)
3. Eligible for any commercialized market authorized anti-CD19 CAR T-cells
4. Performance Status 0 or 1
5. With aggressive large B-cell lymphoma, including:

   * diffuse large B-cell lymphoma
   * Primary mediastinal B-cell lymphoma
   * Any transformed follicular or marginal zone lymphoma
   * high-grade B-cell lymphoma (HGBL) Note: patients with Central Nervous System (CNS) involvement could be included but not patients with primary CNS lymphoma
6. Available biopsy for centralized review
7. With a CAR T-cells indication as soon as 2nd line treatment no later than in 4th line, previously validated by the multidisciplinary tumor board Note: Any treatment performed prior to leukapheresis is considered a line of treatment
8. Total MetabolicTumor Volume (TMTV) > 80 ml, measured by centralized review, on 18FDG-PET (positron emission tomography) done just before starting CAR T-cells procedure (i.e., D-13 +/- 4 days before CAR-T cells infusion)
9. Creatinine clearance (as estimated by Modification of Diet in Renal Disease (MDRD) if > 60-year-old or Cockcroft-Gault if <60yo) >45 mL/min,
10. Adequate hepatic function:

    * aspartate aminotransferase/alanine aminotransferase (ALT/AST) ≤ 3.0 x ULN. (Note: In the case of documented liver involvement by lymphoma, ALT/AST must be ≤ 5.0 x ULN)
    * Serum total bilirubin ≤ 2.0 mg/dL (34 μmol/L) (Note: In the case of Gilbert's syndrome, or documented liver or pancreatic involvement by lymphoma, serum total bilirubin must be ≤ 3.0 mg/dL (51 μmol/L))
11. Patient covered by any social security system (France)
12. Patient who understands and speaks one of the country official languages, unless local regulation authorizes independent translators
13. Contraception:

    * For women of childbearing potential: Agreement to remain abstinent (refrain from heterosexual intercourse) or use two adequate methods of contraception, including at least one method with a failure rate of <1% per year, as soon as consent is signed, during the treatment period (including periods of treatment interruption), and for at least 28 days after the last dose of golcadomide, Women must refrain from donating eggs during this same period.

Exclusion Criteria:

1. History of malignancy other than non-melanoma skin cancer or carcinoma in situ (eg, cervix, bladder, breast) unless disease free for at least 3 years
2. Presence or suspicion of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management; simple urinary tract infection and uncomplicated bacterial pharyngitis are permitted if responding to active treatment and after consultation with the sponsor's medical monitor
3. History of human immunodeficiency virus (HIV) infection or acute or chronic active hepatitis B or C infection; subjects with history of hepatitis infection must have cleared their infection as determined by standard serological and genetic testing per current Infectious Diseases Society of America guidelines or applicable country guidelines
4. Significant pulmonary function impairment and oxygen saturation (SaO2) < 92% on room air
5. Significant cardiovascular disease such as New York Heart Association Class III or IV or Objective Class C or D cardiac disease (see appendix 07)
6. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 6 months of enrollment
7. History of severe immediate hypersensitivity reaction to any of the agents used in this study
8. Current treatment with strong CYP3A4/5 modulators (see appendix 13)
9. Pregnant, planning to become pregnant or lactating Women of Child Bearing Potential
10. Any significant medical conditions, laboratory abnormality or psychiatric illness likely to interfere with participation in this clinical study (according to the investigator's decision)
11. Person deprived of his/her liberty by a judicial or administrative decision
12. Person hospitalized without consent
13. Adult person under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2027-10-20 (Estimated)

PRIMARY OUTCOMES:
Complete metabolic response rate (CMR rate) | 3 months
  efficacy of golcadomide administered post-anti-CD19 CAR T-cell infusion

SECONDARY OUTCOMES:
Objective response rate (ORR) | at 1 month, 3 months, 6 months, 1 year and 2 years, from CAR-T infusion
  incidence of either a complete (CMR) or a partial (PMR) metabolic response per the Lugano Classification (Cheson 2014) as determined by study investigators
Objective response rate (ORR) | at 1 month and 3 months
  determined by imaging central review
Complete response rate (CRR) | at 1 Month, 6 Months, 1 year, and 2 years
  percentage of complete response determined by investigator assessment classification
Duration of response (DR) | 2 years
  time from attainment of PMR or CMR to the date of first documented disease progression/relapse (based on investigator disease assessment (INV)) or death from any cause
Event-free survival (EFS) | 2 years
  the time between CAR T-cells injection and death, disease progression, or start of subsequent new anti-lymphoma therapy including Stem Cell Transplant (SCT)
Progression-free survival (PFS) | 2 years
  time from CAR T-cells injection to the first observation of documented disease progression/relapse (based on investigator disease assessment (INV)) or death
Time To Next anti-Lymphoma Treatment (TTNLT) | 2 years
  from the date of CAR T-cells injection to the date of first documented administration of any new anti-lymphoma treatment
Overall survival (OS) | 2 years
  from date of CAR T-cells injection to the date of death
Incidence of Adverse Events and Serious Adverse events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Catherine THIEBLEMONT, Prof. Dr., Principal Investigator — Hôpital Saint-Louis; Gabriel BRISOU, Prof. Dr., Principal Investigator — Institut Paoli-Calmettes; François-Xavier GROS, Prof. Dr., Principal Investigator — University Hospital, Bordeaux
Locations (13):
- France (13):
  - Hopital Henri Mondor, Créteil
  - Chu Dijon Bourgogne, Dijon
  - Chu de Grenoble, La Tronche
  - Chru de Lille, Lille
  - Institut Paoli Calmettes, Marseille
  - Chu de Montpellier, Montpellier
  - Chu de Nantes, Nantes
  - Hopital Saint-Louis, Paris
  - Chu de Bordeaux, Pessac
  - Chu Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Iuct Oncopole, Toulouse
  - Chu Brabois, Vandœuvre-lès-Nancy